CLINICAL TRIAL: NCT02314741
Title: Peroral Endoscopic Myotomy (POEM) for Esophageal Motility in Patients With a Clinical Diagnosis of Achalasia
Brief Title: Peroral Endoscopic Myotomy (POEM) for Esophageal Motility
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 819130
Record Dates: First submitted 2014-07-17; First posted 2014-12-11 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Achalasia
Keywords: poem; per oral endoscopic myotomy; achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Pyloromyotomy

ARMS (1):
- POEM Treatment Arm (Experimental): Patients treated with the POEM (per-oral endoscopic myotomy) procedure.
  Interventions: Procedure: POEM Procedure

INTERVENTIONS:
Procedure: POEM Procedure — The procedure is performed under anesthesia.The procedure involves endoscopic electrosurgical dissection with an Olympus triangular tip knife.The myotomy is usually ~6cm long & averages 8-10cm. After the myotomy is performed the scope is withdrawn & inserted into the lumen to inspect the mucosa, ensure mucosal integrity & confirm easy passage of the endoscope through the LES consistent with an adequate myotomy. The mucosal entry site is usually 2-3cm long, & is closed with 5-10 endoscopic clips. Patients are hospitalized after procedure for observation.The patient is given IV-nutrition until post-operative day 1. An esophagram is obtained. If no loss of mucosal integrity or leak is noted, a liquid diet is started, which is continued for several days before initiating a solid diet.
  Other Names: POEM; per oral endoscopic myotomy

SUMMARY:
The investigators wish to monitor the adoption of a new, incisionless approach to performing a Heller myotomy for the surgical treatment of achalasia. The method, the Peroral Endoscopic Myotomy (POEM), will provide less-invasive treatment for esophageal achalasia, ideally providing similar if not better outcomes (safety and efficacy) as the Heller myotomy. The investigators hope to enroll 10 patients with a clinical diagnosis of achalasia who meet inclusion criteria.

The POEM procedure has been done in many hospitals without any research associated with it. Dr. Ginsberg, Dr. Chandrasekhara and Dr. Kochman will perform the procedures after being trained. Dr. Ginsberg has personally witnessed the performance of 10 POEM procedures and has performed in a swine model. The PI is credentialed to initiate POEM at HUP with the first case to be proctored by an experienced operator. The PI will then proctor the other adopters. The investigators would like to evaluate the safety of it and the effectiveness of it. The investigators will use their symptom scores and radiology tests pre- and post-POEM to evaluate effectiveness.

DETAILED DESCRIPTION:
An esophageal motility disorder is when muscular contractions become discoordinated or weak and interfere with movement of food down the esophagus. Some esophageal motility disorders persist long enough to cause severe problems requiring surgical intervention. Achalasia, one subtype of esophageal motility disorder that is a rare disease, can be defined by the esophageal sphincter and muscle unable to relax or dilate. Left untreated, symptoms such as difficulty swallowing, regurgitation, heartburn, and chest pain may easily turn into complications such as severe weight loss, malnutrition, coughing, pulmonary infection, pneumonia, and perforation of the esophagus. Diagnosis of esophageal achalasia can be determined by esophageal manometry and/or barium swallow esophagram. Treatment for achalasia includes balloon dilation, botulinum toxin injection and surgical intervention. Balloon dilation is performed by inserting a balloon through the esophageal sphincter, inflating the balloon, disrupting the esophageal muscle. Botox has also been known to successfully relax spastic muscle contractions of achalasia through direct injection into the esophageal muscle. Unfortunately, each alternative to surgical treatment often requires repeated administration to improve the symptoms of achalasia. Traditional treatment of achalasia has included open abdominal or thoracic surgical procedures to cut valve muscles between the esophagus and stomach (Heller Myotomy). Laparoscopic multi-port Heller myotomies have become the preferred approach, requiring 4 smaller abdominal incisions for placement of laparoscope equipment. Results of this laparoscopic technique have proven that although 2/3 of the patient population was successfully treated, a subset of this group still need repeat surgical procedures or balloon dilation. Recently, single-incision laparoscopic Heller myotomies have produced favorable results, with a single umbilical incision preferential to multiple-incision laparoscopy. We propose adoption of a new, incisionless approach to performing a Heller myotomy for the surgical treatment of achalasia. The method, the Peroral Endoscopic Myotomy (POEM) is expected to provide a less-invasive treatment for esophageal achalasia, ideally providing similar if not better outcomes as the Heller myotomy and can be adopted safely and effectively at Penn Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = to 18 years of age
* Clinical diagnosis of achalasia
* A candidate for Heller myotomy
* Esophageal manometry and barium esophogram with findings supportive of achalasia diagnosis
* Women of childbearing potential: negative urine pregnancy test
* Able to undergo general anesthesia
* Willing and able to give informed consent

Exclusion Criteria:

* < 18 years of age
* Pregnancy
* Previous mediastinal or esophageal surgery
* Contraindications for esophagogastroduodenoscopy
* Presence of malignancy
* Coagulopathy (INR 1.5)
* Thrombocytopenia (platelet count < 100K/microliter)
* ASA Score > Class II
* History of mental illness
* Any medical conditions as determined by the PI to be a contraindication to the procedure
* Unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Gather Standardized Data on Patients with Achalasia Who Have Been Treated with the POEM Procedure | About 12 months
  The primary aim of this study is to assess safety and efficacy in the adoption of the POEM procedure compared to the typical Heller Myotomy used for the treatment of achalasia using standardized methods, including esophageal manometry, pre- and post- procedure barium swallow studies, as well as standardized measures of dysphagia symptoms due to achalasia (the Eckart score), and patient's medical records and self-reported symptoms.

SECONDARY OUTCOMES:
Pre-Procedure versus Post-Procedure Barium Swallow Results in POEM Patients | About 6 Months
  Assess POEM procedure's efficacy as defined by improvement of barium swallow study and dysphagia symptoms associated with achalasia. Barium swallow study will compare pre- and post-operative esophageal emptying.
Pre-Procedure Versus Post-Procedure Eckart Score Results in POEM Patients | About 6 Months
  Assess POEM procedure's efficacy as defined by improvement of dysphagia symptoms associated with achalasia. Dysphagia improvement will be assessed using a pre- and post-surgical standardized dysphagia scoring system known as an Eckart Score.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, MD, Principal Investigator — University of Pennsylvania; Gregory G Ginsberg, MD, Principal Investigator — University of Pennsylvania; Gary W Falk, MD, MS, Principal Investigator — University of Pennsylvania; Michael Kochman, MD, Principal Investigator — University of Pennsylvania; David C Metz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States